CLINICAL TRIAL: NCT06225154
Title: Effect of Non-Surgical Periodontal Treatment on Adipokine Levels in Diabetes Mellitus: A Controlled Clinical Trial
Brief Title: Effect of Periodontal Treatment on Adipokine Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Collaborators: University of Turku (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAG-C-DRP-100216-0041
Record Dates: First submitted 2018-02-01; First posted 2024-01-25 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Periodontitis; Diabetes Mellitus, Type 2
Keywords: adipokines; diabetes mellitus; inflammation; periodontitis
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus, Type 2; Diabetes Mellitus; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention (No Intervention): Periodontally healthy subjects with type 2 diabetes mellitus or systemically healthy didn't have an initial periodontal treatment
- Non-surgical periodontal treatment (Experimental): Non-surgical periodontal treatment was performed in a quadrant-wise manner at 1-week intervals for periodontitis patients systemically healthy or with type 2 diabetes mellitus.
  Interventions: Procedure: Non-surgical periodontal treatment

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment — Non-surgical periodontal treatment was performed in a quadrant-wise manner at 1-week intervals.
  Arms: Non-surgical periodontal treatment

SUMMARY:
The present study aimed to determine the effect of non-surgical periodontal treatment (NSPT) on serum and salivary adipokine and interleukin-1β levels in periodontitis patients with or without type 2 Diabetes Mellitus (T2DM).

DETAILED DESCRIPTION:
The present study aimed to determine the effect of non-surgical periodontal treatment (NSPT) on serum and salivary adipokine and interleukin (IL)-1β levels in periodontitis patients with or without type 2 Diabetes Mellitus (T2DM). A total of 80 patients; 20 healthy, 20 T2DM with periodontitis (P), 20 T2DM periodontally healthy, 20 systemically healthy with P were included in this study. At baseline, serum and saliva samples were collected and the whole mouth clinical periodontal parameters were recorded. Periodontitis patients received NSPT in 4 sessions. Clinical parameters were re-measured and samples were re-collected at 1 and 3 months after treatment. Serum and salivary levels of adipokines and IL-1β were analyzed using a flow cytometry-based technique of Lumina® map™. Data were analyzed using appropriate statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus should be diagnosed for ≥1 year and HbA1c level should be at least %6,5
* Periodontitis should be diagnosed for at least 4 teeth with probing depth ≥5 mm with bleeding on probing (BOP) and also radiographic alveolar bone loss should be presence
* Presence of at least 15 teeth

Exclusion Criteria:

* Received antibiotic treatment in the previous 3 months
* Smokers
* Pregnancy and lactation
* Received periodontal treatment in the previous 6 months
* Presence of less than 15 teeth
* Having major diabetic complications

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Serum and Salivary Resistin Levels (pg/ml) | Change between baseline, 1 and 3 months after non-surgical periodontal treatment
  Serum and salivary resistin levels
Serum and Salivary Leptin Levels (pg/ml) | Change baseline, 1 and 3 months after non-surgical periodontal treatment
  Serum and salivary leptin levels
Serum and Salivary Visfatin Levels (pg/ml) | Change baseline, 1 and 3 months after non-surgical periodontal treatment
  Serum and salivary visfatin levels
Serum and saliva IL-1β levels (pg/ml) | Change baseline, 1 and 3 months after non-surgical periodontal treatment
  Serum and salivary IL-1β levels

SECONDARY OUTCOMES:
HbA1c ( %) | Change baseline, 1 and 3 months after non-surgical periodontal treatment
  Glycated Hemoglobin Level %

OTHER OUTCOMES:
Probing Depth (mm) | Change baseline, 1 and 3 months after non-surgical periodontal treatment
  probing depth measured from the gingival margin seldom corresponds to sulcus or pocket depth in mm.
Plaque Index | Change baseline, 1 and 3 months after non-surgical periodontal treatment
  The measurement of the state of oral hygiene by Silness-Löe plaque index is based on recording both soft debris and mineralized deposits on the following teeth. Values 0,1,2 and 3 can be taken. While 0 indicates the least value, 3 indicates the maximum value.
Gingival Index | Change baseline, 1 and 3 months after non-surgical periodontal treatment
  A measure of periodontal disease based on the severity and location of the lesion. Values 0,1,2 and 3 can be taken. While 0 indicates the least value, 3 indicates the maximum value.
Bleeding on Probing (%) | Change baseline, 1 and 3 months after non-surgical periodontal treatment
  Percentage of bleeding sites. Bleeding on probing, often abbreviated BOP, is a sign of inflammation and indicates some sort of destruction and erosion to the lining of the sulcus or the ulceration of sulcular epithelium. The blood comes from lamina propria after the ulceration of the lining.
Clinical Attachment Level (mm) | Change baseline, 1 and 3 months after non-surgical periodontal treatment
  The estimated position of structures that support the tooth as measured with a periodontal probe in mm; provides an estimate of a tooth's stability and of loss of bone support.

CONTACTS AND LOCATIONS:
Overall Officials: Basak Dogan, Prof. Dr., Study Director — Department of Periodontology, Faculty of Dentistry, Marmara University; Yaprak Kalkan, Dt., Principal Investigator — Department of Periodontology, Institute of Health Sciences, Marmara University; Ulvi Kahraman Gürsoy, Assoc. Prof., Study Chair — Department of Periodontology, Institute of Dentistry, Turku University; Mervi Gürsoy, Assoc. Prof., Study Chair — Department of Periodontology, Institute of Dentistry, Turku University; Eija Könönen, Prof. Dr., Study Chair — Department of Periodontology, Institute of Dentistry, Turku University
Locations (2):
- Department of Periodontology, Institute of Dentistry, Turku University, Turku, Lemminkäisenkatu 2, Finland
- Marmara University, Faculty of Dentistry, Department of Periodontology, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Furugen R, Hayashida H, Yamaguchi N, Yoshihara A, Ogawa H, Miyazaki H, Saito T. The relationship between periodontal condition and serum levels of resistin and adiponectin in elderly Japanese. J Periodontal Res. 2008 Oct;43(5):556-62. doi: 10.1111/j.1600-0765.2008.01085.x. Epub 2008 Jun 28. PMID 18565135
- [Background] Gokhale NH, Acharya AB, Patil VS, Trivedi DJ, Setty S, Thakur SL. Resistin levels in gingival crevicular fluid of patients with chronic periodontitis and type 2 diabetes mellitus. J Periodontol. 2014 Apr;85(4):610-7. doi: 10.1902/jop.2013.130092. Epub 2013 Jun 27. PMID 23805816
- [Background] Goncalves TE, Zimmermann GS, Figueiredo LC, Souza Mde C, da Cruz DF, Bastos MF, da Silva HD, Duarte PM. Local and serum levels of adipokines in patients with obesity after periodontal therapy: one-year follow-up. J Clin Periodontol. 2015 May;42(5):431-9. doi: 10.1111/jcpe.12396. Epub 2015 Apr 30. PMID 25858047